CLINICAL TRIAL: NCT03275675
Title: Evaluation of Patients' Satisfaction With the Dispensation of Their Oral Anticancer Treatment in Community Pharmacy: Observational and Transversal Study
Brief Title: Evaluation of Patients' Satisfaction With the Dispensation of Their Oral Anticancer Treatment in Community Pharmacy
Acronym: ORCA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-344; 2017-A01139-44 (Other: 2017-A01139-44)
Record Dates: First submitted 2017-07-31; First posted 2017-09-07 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2018-10

CONDITIONS: Cancer
Keywords: Cancer; Oral chemotherapy; Community Pharmacy; Satisfaction
MeSH Terms: conditions — Neoplasms; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer chemotherapy: This study project is designed to evaluate the satisfaction of patients undergoing oral chemotherapy treated for a cancer and whose treatment is provided by their community pharmacies.
  Interventions: Drug: Oral anticancer medications

INTERVENTIONS:
Drug: Oral anticancer medications — All the oral medications for cancer treatment (hormonal, cytotoxic and targeted therapies)

SUMMARY:
The pharmacist, as a specialist of medications, occupies a strategic position: he participates in a global care of their patients. Dispensation is the pharmaceutical act which associates with the dispensing of medications "the pharmaceutical analysis of the medical prescription if it exists, the possible preparation of the doses to be administered and the provisions of the information and advices necessary for the proper use of medications". The pharmacist ensures that the quality and safety of the dispensation is guaranteed at all times by limiting as far as possible the risks associated with an error in delivery, prescription, drug interactions or undetected contraindications, inadequate dosages or non-compliance with treatment. The longer the patient feels satisfied with the stage of delivery of his treatment, the better his adherence to treatment is, and the less he will encounter poor compliance. Oncology has particularly benefited in recent years from the introduction of numerous drugs with the aim of extending the duration of response in a growing number of indications. Traditionally in oncology, chemotherapy treatments are administered intravenously by trained personnel and rarely managed by the patient at home. Recently, there has been a growing choice of oral formulations, whether for conventional hormonal, anticancer therapies or targeted therapies. These specialties are now widely available in community pharmacies. Oral administration puts the patient at the center of his therapeutic management. He must take his medication alone. Adherence and compliance are therefore particularly important here for an optimal risk-benefit ratio. This study project is designed to evaluate the satisfaction of patients undergoing oral chemotherapy treated for a cancer pathology and whose treatment is provided by their community pharmacies. It also needs to provide information about the reasons for their poor adherence to treatment (personal factors, factors attributable to treatment, factors attributable to the care system). Patients will be recruited and interviewed by contacting several departments of the Clermont-Ferrand University Hospital (CHU de Clermont-Ferrand), who are used to caring for patients with cancerous diseases (hematology, urology, respiratory, gastro-enterology). The data collected in this study may be used for subsequent studies evaluating new management strategies or therapeutic education to improve adherence to patient treatment.

DETAILED DESCRIPTION:
This observational and transversal study will be conducted as a survey by contacting each eligible patients after complete information by the oncologist. After acceptance, the patients will received a postal mail with the questionnaire and a stamped envelope for the return of completed questionnaire. All the completed questionnaires will be recorded in a specific REDCap database for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient (or helping people) receiving oral cancer chemotherapy or oral hormone therapy delivered in community pharmacy for the treatment of cancer
* Non-opposition to participation in the study

Exclusion Criteria:

* Patient unable to understand or respond to questionnaires
* Age < 18
* Legal incapacity (person deprived of liberty or under guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study project is designed to evaluate the satisfaction of patients undergoing oral chemotherapy treated for a cancer pathology and whose treatment is provided by their community pharmacies. It also needs to provide information about the reasons for their poor adherence to treatment (personal factors, factors attributable to treatment, factors attributable to the care system).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Assessment of patients' satisfaction with the dispensation of their oral anticancer treatments in community pharmacy | at day 1
  (visual analogic scale 0-100)

SECONDARY OUTCOMES:
Assessment of patients' satisfaction based on Quality of Information Provided by Oncologists and Pharmacists | at day 1
  (visual analogic scale 0-100)
Assessment of patients' satisfaction based on type of cancer | at day 1
Assessment of patients' satisfaction based on type of treatment received | at day 1
Assessment of patients' satisfaction based on number of medications taken per day | at day 1
Assessment of patients' satisfaction based on patient characteristics | at day 1
  age, gender, professional status, marital status, level of study

CONTACTS AND LOCATIONS:
Overall Officials: David BALAYSSAC, PhD, PharmD, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France